CLINICAL TRIAL: NCT01399073
Title: Virtual Reality for Neglect Diagnostics
Acronym: KMS-Neglect
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Median Klinik Kladow (Unknown); Freie Universität Berlin (Other); Berlin Center for Advanced Neuroimaging (Unknown); Humboldt-Universität zu Berlin (Other); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. Andreas Meisel, Charite University, Berlin, Germany
Other Study IDs: KMS-Neglect
Record Dates: First submitted 2011-07-08; First posted 2011-07-21 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Spatial Neglect; Stroke
Keywords: stroke; neglect; hemianopsia; virtual reality
MeSH Terms: conditions — Stroke; Hemianopsia | interventions — Paper

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with Neglect
  Interventions: Behavioral: virtual reality setup; Behavioral: paper and pencil tests; Other: c-mri
- Patients with Hemianopsia
  Interventions: Behavioral: virtual reality setup; Behavioral: paper and pencil tests; Other: c-mri
- Healthy age-matched controls
  Interventions: Behavioral: virtual reality setup; Behavioral: paper and pencil tests; Other: c-mri

INTERVENTIONS:
Behavioral: virtual reality setup — testing for neglect in a virtual reality setup
Behavioral: paper and pencil tests — testing for neglect with the classical paper-and-pencil tests
Other: c-mri — structural and functional (resting state) imaging

SUMMARY:
Compared to the classical "paper and pencil"-tests, testing patients in our virtual reality setup might have a higher sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria for neglect patients:

* age ≥18 and <80 years
* first stroke
* neglect symptoms
* no hemianopsia symptoms
* consent given by the patient

Inclusion Criteria for hemianopsia patients:

* age ≥18 and <80 years
* first stroke
* no neglect symptoms
* hemianopsia symptoms
* consent given by the patient

Inclusion Criteria for Controls:

* age ≥18 and <80 years
* no neurological deficits
* informed consent

Exclusion Criteria (for all groups):

* language comprehension deficits
* motor deficits of the upper extremities
* cognitive impairments (MMSE <20 or SKT >15 or DEMTEC >12)
* depression
* seizure disorders
* claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute (< 2 wks after stroke), subacute (2 wks- 3 months after stroke)or chronic (3- 24 months after stroke)stroke with neglect or hemianopsia.
  Healthy, age-matched controls.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Feasibility | within the first 2 years after stroke
  Feasibility of the use of a virtual reality setup in the diagnostics of neglect

SECONDARY OUTCOMES:
Sensitivity and Specificity | within the first 2 years after stroke
  The diagnostics of neglect via a virtual reality setup is more sensitive and more specific than the standard diagnostics via "paper-and-pencil" Tests
mri (functional (resting state) and structural imaging | within the first 2 years after stroke
  We hypothesize that there are connectivity-based differences in the different stages of neglect and anatomical and functional connectivity correlates with respect to behavioural impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, MD, Principal Investigator — Charite University (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center NCRC)
Locations (1):
- Charité University Medicine, Berlin, Germany

REFERENCES:
- [Result] Ulm L, Wohlrapp D, Meinzer M, Steinicke R, Schatz A, Denzler P, Klehmet J, Dohle C, Niedeggen M, Meisel A, Winter Y. A circle-monitor for computerised assessment of visual neglect in peripersonal space. PLoS One. 2013 Dec 12;8(12):e82892. doi: 10.1371/journal.pone.0082892. eCollection 2013. PMID 24349387